CLINICAL TRIAL: NCT03329326
Title: Comparison of Prosthetic Assessment Tools and Factors Influencing the Outcome
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University Medical Center Goettingen (Other); Lund University (Other); Örebro University, Sweden (Other); Helsinki University Central Hospital (Other); BG Trauma Center Ludwigshafen (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Agnes Sturma, BSc, MSc, Medical University of Vienna
Other Study IDs: 1713/2016
Record Dates: First submitted 2017-10-25; First posted 2017-11-01 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Amputation; Prosthesis User
Keywords: standardized test; prosthesis; upper limb amputation; rehabilitation outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional tests and self-reported questionnaires — In this observational study no intervention is initiated. Patients included are only assessed with the non-invasive tests described earlier.

SUMMARY:
Background and rational:

A large number of instruments exists to assess upper limb prosthetic function. However, they differ substantially in terms of psychometric properties and content. Furthermore, there is no "gold standard" and nearly every single center uses a unique set of instruments. This fact prevents the linking of the commonly small (due to the limited number of patients in each center) data sets of different centers and makes comparisons between different fittings or treatment protocols difficult. To generate accepted evidence, we need large data sets with similar outcomes. With remarkable progress made in prosthetic research and rehabilitation in the recent years, the need to evaluate the impact of this intervention on daily life, including productivity, self-care and leisure becomes increasingly relevant. Moreover, self-reported instruments and observation-based instruments exist, but there is a lack of data if, for example, the self-reported instrument (which is easier and less health-professional's-time-consuming to perform) could "replace" a performance or observation-based instrument.

Therefore, the aim of this study is to determine psychometric properties of the existing instruments (SHAP, DASH, SF-36 and ACMC) in a large international data set, to explore possible linkage between self-reported and performance or observation-based instruments and to develop state-of-the art recommendations/points to consider on how to assess functioning in prosthetic care.

DETAILED DESCRIPTION:
Background and rational:

A large number of instruments exists to assess upper limb prosthetic function. However, they differ substantially in terms of psychometric properties and content. Furthermore, there is no "gold standard" and nearly every single center uses a unique set of instruments. This fact prevents the linking of the commonly small (due to the limited number of patients in each center) data sets of different centers and makes comparisons between different fittings or treatment protocols difficult. To generate accepted evidence, we need large data sets with similar outcomes. With remarkable progress made in prosthetic research and rehabilitation in the recent years, the need to evaluate the impact of this intervention on daily life, including productivity, self-care and leisure becomes increasingly relevant. Moreover, self-reported instruments and observation-based instruments exist, but there is a lack of data if, for example, the self-reported instrument (which is easier and less health-professional's-time-consuming to perform) could "replace" a performance or observation-based instrument.

Therefore, the aim of this study is to determine psychometric properties of the existing instruments in a large international data set, to explore possible linkage between self-reported and performance or observation-based instruments and to develop state-of-the art recommendations/points to consider on how to assess functioning in prosthetic care. Projects exploring outcome assessments should have a broad basis and target different patient populations. To be able to generalize the outcome of the study for the European population, this study is planned as a multi-centre study. Also, having a sufficient number of subjects to calculate statistical relationships is otherwise not possible due the limited number of patients being treated at most centers.

Included patients:

* age: 16-85 years
* major uni-lateral amputation of the upper extremity (includes amputation of the hand, forearm, upper arm and at shoulder level)
* normal hand function of the other side (in case of doubt: SHAP score ≥ 95)
* no major neurologic or untreated psychological disorders
* fitted with an active prosthesis (myo, body-powered or hybrid) for at least 6 months

Used Assessments:

* Southampton Hand Assessment Procedure (SHAP): The Southampton Hand Assessment Procedure (SHAP) is a clinically validated hand function test developed to assess the effectiveness of upper limb prostheses. The SHAP is made up of 6 abstract objects and 14 Activities of Daily Living (ADL). Each task is timed by the participant, so there is no interference or reliability on the reaction times of the observer or clinician. The SHAP Index of Function score is used for comparison, which is a number that provides an overall assessment of hand function. SHAP scores do not plateau at 100, instead scores greater than 100 can be achieved if a participant is exceptionally quick at a given task or series of tasks. Scores less than 100 are an indication of how impaired a participant's hand function is. In general, scores between 95 and 105 are considered normal.
* Disabilities of Arm, Shoulder and Hand Questionnaire (DASH): The DASH is a questionnaire, where patients are asked to rate their (bimanual) performance in daily life. It has been validated for use in patients with musculoskeletal diseases and injuries to the arm. A score of 100 indicates the worst and 0 indicates the best hand function.
* Short Form -36 Quality of Life Questionnaire (SF-36): We will use the SF-36 Health Survey 4-week recall version. The questionnaire addresses eight independent subscales: physical functioning, physical role functioning, bodily pain, general health, vitality, social role functioning, emotional role functioning, and mental health. Each subscale ranges from 0 to 100. Based on the subscales, two superior physical and mental component summary scales can be identified. These have mean values of 50 and an SD of 10. A (German) patient with a psychological sum scale of 65 exhibits above average mental health compared with age-matched and sex-matched Germans.
* Open questions concerning demographic data and prosthesis-related questions (~15): These questions are used to determine further factors that may influence the outcome of self-rated and performance-based tests. They include factors that are already known to influence upper extremity function or perceived disability (e.g rate at amputation, time since amputation, dominant vs. non-dominant hand), as well as factors that may influence the outcome, but were not studied before in sufficient detail (as living alone).
* Assessment of Capacity of Myoelectric control (ACMC): The "Assessment of Capacity for Myoelectric Control" (ACMC) is an observational assessment developed to assess the ability of a prosthesis user to control a myoelectric prosthetic hand. Each item in the ACMC is an observable prosthetic hand movement, such as timing during grasping, or an observable prosthetic hand movement in relation to other body parts, such as uses the prosthesis over the shoulder. The ACMC assesses how skillful a prosthesis hand user performs different prosthetic hand movements when performing a bimanual activity. To perform the ACMC, a two-day training course is required. As not all participating centres have trained professionals, the use of the ACMC is not mandatory.

Data collection:

* As this is a cross-sectional study, all assessments are performed at one point in time (maximum of 2 months in between the different assessments).
* The participating centers can collect all data by themselves and send (anonymized) data sets to the Medical University of Vienna (MUV). Otherwise, they can invite patients and an experienced physical therapist from MUV will visit the center to do the assessments.

Research questions and statistical considerations:

1. To determine psychometric properties of the existing instruments in a large international data set --> Linkage of data from different centers, psychometric properties; planned analyses: descriptive statistics, correlation, principal components analyses and Rasch analyses
2. To explore possible linkage between self-reported and performance or observation-based instruments. planned analyses: Regression analyses
3. To develop state-of-the art points to consider on how to assess functioning in prosthetic care

Anticipated sample size:

The aim of this study is to get a (representative) sample of the European prosthesis using population, which presents the major the reason for the multi-centre study design. The planned sample size is 100-200 amputees fitted with an active prosthesis. This number should alow proper statistic calculations of the influence of the co-variants, but also be feasible with the number of centres participating.

ELIGIBILITY:
Inclusion Criteria:

* age: 16-85 years
* major uni-lateral amputation of the upper extremity
* normal hand function of the other side (in case of doubt: SHAP score ≥ 95)
* fitted with an active prosthesis for at least 6 months
* gives informed consent

Exclusion Criteria:

* major neurologic or untreated psychological disorders

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes upper-limb amputees who are fitted with an acitve prosthesis. it is intented to have a diverse sample concerning age, gender, time since amputation,...
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Southampton Hand Assessement Procedure | 1 day
  standardized test for prosthetic function
Disabilities of Arm Shoulder and Hand | 1 day
  questionnaire for hand function

SECONDARY OUTCOMES:
Assessment of the Capacity of Myoelectric Control | 1 day
  standardized test for prosthetic function
Short Form 36 | 1 day
  questionnaire for health-related quality of life

OTHER OUTCOMES:
Time since amputation [years] | 1 day
  Patients are asked for how long they have been an amputee.
Time since fitting [years] | 1 day
  Patients are asked for how long they are fitted with an active prosthesis.
Living alone [yes/no] | 1 day
  Patients are asked, if they live alone in their household.
dominant hand amputated [yes/no] | 1 day
  Patients are asked if the amputated side was their dominant one before amputation.
gender [male/female/other] | 1 day
  Patients are asked about their gender.
having children [yes/no] | 1 day
  Patients are asked, if they have children.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes BM Sturma, BSc. MSc., Principal Investigator — Medical University of Vienna
Locations (7):
- Medical University of Vienna, Vienna, Austria
- Helsiniki University Central Hospital, Helsinki, Helsiniki, Finland
- Germany (2):
  - University Medical Center Goettingen, Goettigen, Lower Saxony
  - BG Trauma Center Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate
- Sykehuset Innlandet HF, Ottestad, Norway
- Sweden (2):
  - Lund University, Lund, Skåne County
  - Örebro University, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be discussed within the group of participating centres upon specific request.

REFERENCES:
- See also: Further information about the DASH — http://www.dash.iwh.on.ca/
- See also: Further information about the SHAP — http://www.shap.ecs.soton.ac.uk/
- See also: Further information about the ACMC — http://acmc.se/